CLINICAL TRIAL: NCT04776811
Title: Evaluation of Accuracy of Guardian Sensor 3 in Diabetes Patients on Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: Elaine Chow (Other)
Collaborators: Medtronic Diabetes (Industry)
Responsible Party: Sponsor-Investigator, Elaine Chow, Clinical Assistant Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: PDGS3
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus (Diagnosis); End Stage Renal Disease; Dialysis
MeSH Terms: conditions — Diabetes Mellitus; Disease; Kidney Failure, Chronic | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous glucose monitoring system — Medtronic Guardian Connect with Guardian Sensor 3

SUMMARY:
Assessment of performance (precision and accuracy) of Guardian Sensor™ 3 as compared with a gold standard reference laboratory method (YSI glucose) in diabetes patients on peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetes mellitus diagnosed for at least 3 months
2. On continuous ambulatory peritoneal dialysis (CAPD) for at least 3 months
3. Male or female age ≥ 18 years old and ≤ 75 year old.
4. Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study.
5. Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) frequency of clinic visits and use of pre-specified glucose monitoring devices.
6. Willingness to abstain from swimming during their participation in the measurement phase.
7. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a good study candidate.
8. Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

1. Poorly controlled diabetes mellitus with HbA1c>11%
2. Peritonitis within 1 month
3. On icodextrin PD solutions
4. Planned for switching to hemodialysis or living donor transplant in future 3 months
5. Currently pregnant, as demonstrated by a positive pregnancy test at screening
6. Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
7. Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
8. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
9. Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
10. Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study.
11. Blood donation of more than 500 ml within the last three months
12. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.

13 Has a MRI scan, CT scan, or diathermy scheduled during the proposed study participation.

14. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

15. Women of reproductive potential who are unwilling to adopt contraceptive measures during the study period 16. Patients with history of pacemaker and prosthesis implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes patients on continuous ambulatory peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative difference (MARD) | 5 minutes
  MARD of sensor versus YSI glucose

SECONDARY OUTCOMES:
Median absolute relative difference (MedARD) | 5 minutes
  MedARD of sensor versus YSI glucose
Consensus Error grid analysis | 5 minutes
  % sensor values in regions A and B
Percent accuracy | 5 minutes
  System readings within 15%, 20%, 30%, 40% and greater than 40% of YSI values
Hypoglycemia detection rates | 15 minutes
  True and false hypoglycemia notification rate, correct and missed hypoglycemia detection rate
Hyperglycemia detection rates | 15 minutes
  True and false hyperglycemia notification rate, correct and missed hyperglycemia detection rates
User satisfaction | 2 weeks
  Diabetes Satisfaction Treatment Questionnaire score
Correlation between CGM metrics, HbA1c and fructosamine | 2 weeks
  Correlation between CGM metrics, HbA1c and fructosamine

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, PhD, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Elaine Chow, Hong Kong, None Selected, China

IPD SHARING:
Plan to Share IPD: No